CLINICAL TRIAL: NCT07061106
Title: Comparison of Otago and Kitchen Sink Balance Exercises on Strength, Fall Risk and Functional Mobility on Elderly.
Brief Title: Otago and Kitchen Sink Balance Exercises on Strength, Fall Risk and Functional Mobility on Elderly.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Asiya Naeem
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Fall Risk, Fall Prevention
Keywords: Otago, Kitchen Sink, fall risk, strength, functional mobility, Elderly

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Otago exercise program (Experimental): Group will receive intervention of 45 minutes per session, 3 times a week, and for a total of 8 weeks (24 sessions).
  Interventions: Other: Otago exercise program
- Kitchen Sink Balance Exercises (Active Comparator): Group will receive intervention of 45 minutes per session, 3 times a week, and for a total of 8 weeks (24 sessions).
  Interventions: Other: Kitchen Sink Balance Exercises

INTERVENTIONS:
Other: Otago exercise program — Study will be conducted after the approval of Ethical review board. After the initial evaluation will be done on participants underlying eligibility criteria. Intervention Group A received Otago Exercise Program and will receive intervention of 45 minutes per session, 3 times a week, and for a total of 8 weeks (24 sessions). The Otago Exercise Program is a fall prevention well designed program for older adults. It includes 17 strength and balance exercises and a walking program, which are typically performed three times a week and helps to prevent falls in older adults by strengthening muscles and improving balance. In this study, modified form of Otago would be used that focuses on balance and strengthening exercises.
  Arms: Otago exercise program
Other: Kitchen Sink Balance Exercises — Study will be conducted after the approval of Ethical review board. After the initial evaluation will be done on participants underlying eligibility criteria. Intervention Group B received Kitchen Sink Balance Exercises and will receive intervention of 45 minutes per session, 3 times a week, and for a total of 8 weeks (24 sessions). Kitchen sink balance exercises are beneficial for improving overall Individual's stability, strength, and coordination. These exercises can be easily integrated into daily routine and it also providing a practical way to enhance balance and overall fitness.
  Arms: Kitchen Sink Balance Exercises

SUMMARY:
The objective of the study is to determine the comparative effects of Otago Exercise Program and Kitchen Sink Balance Exercises on strength, fall risk and functional mobility on elderly. This study would include total 56 participants which would be divided into two groups, 28 each. Convenience Sampling will be used and randomly assigned into two groups through sealed envelope method. Intervention Group A received Otago Exercise Program and Group B received Kitchen Sink Balance Exercises. Both groups received intervention for 45 minutes per session, 3 times a week, and for a total of 8 weeks. Assessment was done at the baseline, after 4 weeks and after 8 weeks.

DETAILED DESCRIPTION:
Issues with balance are a leading cause of falls and are associated with enhanced fear of falling and also reduced the confidence in balance. The decline in balance with age is a complex process involving the body's systems like visual, vestibular, and musculoskeletal systems that working together to maintain the posture stability. Exercise is commonly recommended to enhance balance, muscle strength, and mobility in older individuals. The Otago Exercise Program (OEP) is a proven and well developed intervention that integrates balance and strengthening exercises with walking that tailored for older adults living independently in the community. Exercises at the Kitchen Sink balance program is also effective exercise program designed to prevent falls among older adults and helps to improve balance, increases strength, endurance and flexibility in elderly population. Therefore, we conduct this research to find out the comparative effects of Otago Exercise Program and Kitchen Sink Balance Exercises on strength, fall risk and functional mobility on elderly. It could provide valuable insights into the effectiveness of these interventions for improving balance and reducing risk of falls in elderly population. This research could also help to identify the most effective rehabilitation strategies for elderly individuals with balance problems, ultimately improving their quality of life and reducing healthcare costs associated with falls and balance-related injuries.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 65 and older.
* Both males and females.
* Individuals have a score on BBS (21-40)
* Willingness to participate

Exclusion Criteria:

* Individuals with Severe Cognitive Impairment that would impede understanding and following exercise instructions.
* Individuals having Conditions that contraindicate exercise. (e.g. severe cardiovascular disease)
* Individuals with psychiatric disorders and malignancies.
* Individuals Aged less than 65 years.
* Individuals who are already involve in other balance training program.
* Individuals who are not willing.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | 8 weeks
  BBS is used for assessment of balance and is considered as a gold standard. It consist of 14 simple task and it takes almost 15-20 minutes to complete. Its 0-4 grading scale where 0 means unable and 4 means independent. Overall score is 56 having interpretation of <20 indicative of wheel chair user, >20-<40 walking with assistance and >40-56 showing independency of patient. On BBS cut-off score of 40 points provided optimal sensitivity of 0.82 and specificity of 0.67.
Short Physical Performance Battery Score Tool (SPPB) | 8 weeks
  SPPB is a group of objective assessment tools for balance, lower extremity strength, and functional mobility in older adults (>65 years of age). The test includes three different domains like walking, sit-to-stand and balance to assess individual's functional mobility. The scoring of this tool range from 0 (worst performance) to 12 (best performance).

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Azhar, MS-NMPT, Principal Investigator — Riphah International University
Locations (1):
- Najjat Trust, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No